CLINICAL TRIAL: NCT01229111
Title: A Phase 2 Study of AZD2171 (Cediranib) With Modified FOLFOX6 in Patients With Advanced Biliary Cancers
Brief Title: Cediranib Maleate and Combination Chemotherapy in Treating Patients With Advanced Biliary Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Drug Supply
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02535; NCI-2011-02535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687126; CASE 9209 (Other: Case Comprehensive Cancer Center); 8323 (Other: CTEP); N01CM00070 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Adult Primary Cholangiocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Localized Unresectable Adult Primary Liver Cancer; Periampullary Adenocarcinoma; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — cediranib; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cediranib maleate and modified FOLFOX) (Experimental): Patients receive cediranib maleate PO QD on days 1-14 and modified FOLFOX6 comprising oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1.
  Interventions: Drug: cediranib maleate; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil

INTERVENTIONS:
Drug: cediranib maleate — Given PO
  Other Names: AZD2171; Recentin
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
This phase II trial is studying how well giving cediranib maleate together with combination chemotherapy works in treating patients with advanced biliary cancers. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cediranib maleate together with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate to AZD2171 (cediranib maleate) and modified folinic acid-fluorouracil-oxaliplatin-6 regimen (FOLFOX 6) in subjects with advanced biliary cancers.

SECONDARY OBJECTIVES:

I. To determine overall assessment of toxicity of AZD2171 and modified FOLFOX6. II. To determine the progression-free survival of subjects with advanced biliary cancers treated with AZD2171 and modified FOLFOX6.

III. To determine overall survival of subjects with advanced biliary cancers treated with AZD2171 and modified FOLFOX6.

OUTLINE:

Patients receive cediranib maleate orally (PO) once daily (QD) on days 1-14 and modified FOLFOX6 comprising oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathological or cytopathological diagnosis of advanced biliary carcinoma (gallbladder cancer, cholangiocarcinoma, ampullary cancer) not amenable to conventional surgical approach are eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan
* No patients with untreated brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Life expectancy of greater than 12 weeks
* White blood cell (WBC)/leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 3 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 times institutional upper limit of normal
* Creatinine within normal institutional limits OR calculated creatinine clearance ≥ 60 mL/min
* No patients with proteinuria not meeting the criteria below; urine sample must be tested by urine protein:creatinine (UPC) ratio or by urinalysis method within 1 week of starting study treatment; depending upon the testing method used, the following criteria must be met:

  * UPC ratio must be < 1.0; if UPC ratio is ≥ 1.0, a 24-hour urine specimen must be collected and must demonstrate < 1 g of protein
  * Urinalysis must indicate 0-1+ protein; if urinalysis reading is ≥ 2+, a 24-hour urine specimen must be collected and must demonstrate < 1 g of protein
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use adequate contraception (hormonal or barrier method of birth control; abstinence) before and during study treatment

  * Acceptable contraception includes abstinence, oral contraceptives, intra-uterine device (IUD), diaphragm, Norplant, approved hormone injections, condoms, or documentation of medical sterilization
* Patients with evidence of heart disease must be New York Heart Association (NYHA) Class I or II

  * NYHA Class II patients controlled with treatment are considered at increased risk for compromised left ventricular ejection fraction (LVEF) and will undergo increased cardiac monitoring
* No patients with other active invasive cancers except nonmelanoma skin cancer or carcinoma in-situ of the cervix

  * History of prior cancer is allowed as long as there has been no evidence of disease within the past 5 years
* No patients with mean corrected QT interval (QTc) > 480 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome
* No patients with uncontrolled hypertension defined as systolic blood pressure (BP) ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg, with or without anti-hypertensive medication or history of hypertensive crisis or hypertensive encephalopathy

  * Patients with initial BP elevations are eligible once their BP is controlled to above parameters
* No patients with uncontrolled intercurrent illness including, but not limited to:

  * Hypertension (> 140/90 mm Hg)
  * Chronic or active infection requiring chronic suppressive antibiotics
  * History of or symptomatic congestive heart failure requiring chronic medical therapy
  * NYHA class III or IV heart disease
  * Unstable angina pectoris within 180 days prior to starting study treatment
  * Myocardial infarction within 180 days prior to study treatment
  * Gastroduodenal ulcer(s) determined by endoscopy to be active within 180 days prior to study treatment
  * Serious or non-healing wound, skin ulcers, or bone fracture
  * Any significant bleeding that is not related to the primary tumor within 180 days prior to study treatment
  * Known bleeding diathesis or coagulopathy
  * Paresthesias, peripheral sensory neuropathy > gr. 1 per Common Terminology Criteria for Adverse Events (CTCAE) v.4, or peripheral motor neuropathy ≥ gr. 2 per CTCAE v.4
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No patients with history of transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 180 days prior to study treatment, symptomatic peripheral ischemia; history of arterial thrombotic event within 180 days prior to study treatment; gastrointestinal (GI) perforation within 180 days prior to study treatment
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who are chemotherapy naive unless chemotherapy was given as adjuvant post-surgical treatment and at least 6 months have elapsed since adjuvant chemotherapy
* No patients who have had major surgical procedures, open biopsies, or significant traumatic injury within 28 days prior to study treatment
* Chemotherapy for prior cancer is permitted
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or PK of AZD2171 will be determined following review of their case by the Principal Investigator

  * Efforts should be made to switch patients with brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial within the past 30 days
* Patients may not be receiving any medication that may markedly affect renal function (e.g., vancomycin, amphotericin, pentamidine)
* Patients may not be receiving therapeutic doses of Coumadin or equivalent
* No patients requiring drugs with proarrhythmic potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, Principal Investigator — Case Comprehensive Cancer Center
Locations (7):
- United States (7):
  - Seidman Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Ireland Cancer Center Landerbrook Health Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from hospitals in Cleveland and Columbus, Ohio from October 2010 through February 2013.
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Started | 14
Completed | 13
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All patients who signed consent.
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Number analyzed (Participants) | 14
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 1
  50-59 years | 3
  60-69 years | 8
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: The Response Rate of Patients Evaluated Using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: The number of patients with a Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions); Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 3 years
Population: Patients that were evaluable
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Number analyzed (Participants) | 11
participants
  Partial Response (PR) | 4
  Stable Disease (SD) | 6
  Progressive Disease (PD) | 1

2. Secondary Outcome: Tabulation of the Toxicity Profile of the Combination Therapy
Description: Number of patients that experienced >/= grade 3 treatment related toxicities (definite, probable, possible).
Time Frame: Up to 3 years
Population: All patients that received treatment drug
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Number analyzed (Participants) | 13
participants | 11

3. Secondary Outcome: Progression Free Survival
Description: Time in months that evaluable subjects survived progression free
Time Frame: Up to 3 years
Population: Patients that were evaluable for response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Number analyzed (Participants) | 13
Months | 14.4 [3 to 22.5]

4. Secondary Outcome: Estimation of Overall Survival
Description: Time of overall response
Time Frame: Up to 3 years
Population: Patients that received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Number analyzed (Participants) | 13
Months | 19.2 [3 to 31.3]

5. Secondary Outcome: Identification of Factors That Predict Survival
Description: Factors that predict survival will be identified by Cox model or extended Cox model.
Time Frame: Up to three years
Population: Statistically, due to the small sample size, analysis could not be done
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from start of treatment until resolved for about 3 years.
Arm/Group | Treatment (Cediranib Maleate and Modified FOLFOX)
Serious Adverse Events (participants affected / at risk) | 11/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate and Modified FOLFOX) (N=13)
Anemia (Blood and lymphatic system disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal hemorrage (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal Obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Death (General disorders) | 2
Fatigue (General disorders) | 1
Biliary Tract infection (Infections and infestations) | 1
Catheter related infection (Injury, poisoning and procedural complications) | 2
Skin Infection (Infections and infestations) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Disease Progression
Altered mental status (Nervous system disorders) | 1
Confusion (Pregnancy, puerperium and perinatal conditions) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Abscess (Gastrointestinal disorders) | 1
Fibrile Neutropenia (Blood and lymphatic system disorders) | 1
Lung Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate and Modified FOLFOX) (N=13)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 11
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 13
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Anal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 11
Anxiety (Psychiatric disorders) | 6
Aortic valve disease (Cardiac disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 10
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Biliary tract infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 5
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Catheter related infection (Cardiac disorders) | 2
Chest pain - cardiac (Psychiatric disorders) | 1
Confusion (Gastrointestinal disorders) | 1
Constipation (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Investigations) | 2
Creatinine increased (Metabolism and nutrition disorders) | 2
Dehydration (Psychiatric disorders) | 3
Depression (Gastrointestinal disorders) | 4
Diarrhea (Nervous system disorders) | 8
Dizziness (Gastrointestinal disorders) | 8
Dry mouth (Skin and subcutaneous tissue disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Edema limbs (General disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flushing (Vascular disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 3
Hemoglobin increased (Investigations) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Hot flashes (Vascular disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Infections and infestations - thrush (Infections and infestations) | 3
Insomnia (Psychiatric disorders) | 10
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Investigations) | 6
elevated LDH (Investigations) | 4
Mucositis oral (Gastrointestinal disorders) | 8
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - cold sensitivity (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 9
Non-cardiac chest pain (General disorders) | 2
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 11
Platelet count decreased (Investigations) | 12
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Skin infection (Infections and infestations) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Urinary tract infection (Infections and infestations) | 3
Urinary tract pain (Renal and urinary disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 10
Wound dehiscence (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less